CLINICAL TRIAL: NCT06902883
Title: Study on the Effectiveness and Comfort of Innovative Solutions for the Internal Transport of Patients in Wheelchairs in a Hospital Setting
Acronym: PreDoPTI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-A00077-40/1; 2024/3801 (Other: CSET number (Gustave Roussy ID))
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Hospitalized Patient

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wheelchair test 1 (Experimental): Patient will test experimental wheelchair during outward journey and standard wheelchair during return journey
  Interventions: Device: Serum holder connected to the wheelchair; Device: wheelchair seat
- Wheelchair test 2 (Experimental): Patient will test standard wheelchair during outward journey and experimental wheelchair during return journey
  Interventions: Device: Serum holder connected to the wheelchair; Device: wheelchair seat

INTERVENTIONS:
Device: Serum holder connected to the wheelchair — Serum holder connected to the wheelchair
Device: wheelchair seat — wheelchair seat

SUMMARY:
In 2006, 2012, and 2018, under the auspices of the Pain Control Committee, Gustave Roussy stretcher-bearers conducted studies on patient pain caused by internal transport (stretchers). The first study showed that this pain is primarily experienced by patients initially in pain, and that risk factors include crossing elevator landings and threshold bars, handling, and prolonged waiting times.

A progress plan was developed, and since 2006, improvement initiatives have been regularly implemented. Their effectiveness has been evaluated by patients and the professionals involved (departure department, carrier, and arrival department).

Stretcher-bearing software was purchased following the original study; scheduling has been streamlined, journeys are transmitted to stretcher-bearers via smartphones, and transport times are calculated and analyzed. In 2019, a prototype for connecting patients' IV poles to wheelchairs was developed and tested, thanks to a collaboration between technical services, stretcher-bearers, and the Bureau of Biostatistics and Epidemiology. The time spent by stretcher-bearers transferring infusion sets and other syringe pumps from the patient's IV pole to the wheelchair's pole on the way out, and vice versa on the way back to the room, has been eliminated. The hypothesis is that this elimination would reduce travel times and could have an indirect impact on reducing pain.

Wheelchair comfort has been continually improved since 2006: the front casters were replaced with softer and thicker ones, the rear wheels with soft wheels and then with pneumatic tires; the backrests were replaced with a memory foam model, and the seats with an "ultra-comfort" model. These improvements contribute to better pain management during transport and an improved patient experience. Wheelchair comfort could be further improved by replacing the seats with high-quality "Bultex" models.

In 2022, 33,800 patients were transported in wheelchairs (round trip, one-way or one-way), representing 35% of annual transports. Technical developments and improvements in wheelchair comfort could contribute to reducing pain caused by internal transport.

Primary Objective To evaluate the effect of two interventions (a system for connecting the IV pole to the wheelchair and a new seat) during the internal transport of cancer patients being treated at Gustave Roussy:

Intervention 1: To evaluate the impact of using the IV pole connection system on reducing the duration of wheelchair transport for patients receiving infusions; Intervention 2: To evaluate patient preference for the comfort of a wheelchair seat.

Secondary Objective To evaluate pain in transported patients (before/after)

ELIGIBILITY:
Inclusion Criteria:

* Informed patient and signed informed consent
* Age equal or greater than 18
* Speak and read french
* For serum holder connected to wheelchair only : patients with multiple infusion devices and transported in wheelchair
* For wheelchair seat : patients transported in wheelchair from hospitalized unit to radiology department

Exclusion Criteria:

* disoriented or confused patient
* Patients under judicial protection (curatorship, tutorship) and/or deprived of freedom
* pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2025-06-16 (Actual); Primary Completion 2025-08-19 (Actual); Study Completion 2025-08-19 (Actual)

PRIMARY OUTCOMES:
Period of transportation | 1 day
  Unit of measurement: minute
Comfort of the wheelchair | 1 day
  Comfort of the wheelchair evaluated according to satisfaction scale from 0 (uncomfortable) to 10 (very comfortable)

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, France

IPD SHARING:
Plan to Share IPD: No